CLINICAL TRIAL: NCT01973660
Title: PAMELA: PAM50 HER2-enriched Phenotype as a Predictor of Early Response to Neoadjuvant Lapatinib Plus Trastuzumab in Stage I to IIIA HER2-positive Breast Cancer
Brief Title: PAM50 HER2-enriched Phenotype as a Predictor of Response to Dual HER2 Blockade in HER2-positive Early Breast Cancer
Acronym: PAMELA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-1114; 2013-001036-22 (EudraCT Number)
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: Human Epidermal Growth Factor Receptor 2; HER2; HER2 positive; PAM50; lapatinib; trastuzumab; dual HER2 blockade; neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab; Letrozole; Tamoxifen; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual HER2 blockade (Experimental): For a total of 18 weeks, HR-negative patients will be given dual blockade consisting of daily lapatinib at 1000 mg and trastuzumab at a loading dose of 8 mg/kg, followed by 6 mg/kg every 3 weeks.
  Interventions: Drug: Lapatinib; Drug: Trastuzumab; Drug: Paclitaxel
- Dual HER2 blockade plus endocrine therapy (Experimental): For a total of 18 weeks, HR-positive patients will be given letrozole (2.5 mg daily) or tamoxifen (20 mg daily) with concurrent dual blockade consisting of daily lapatinib at 1000 mg and trastuzumab at a loading dose of 8 mg/kg, followed by 6 mg/kg every 3 weeks.
  Interventions: Drug: Lapatinib; Drug: Trastuzumab; Drug: Endocrine Therapy; Drug: Paclitaxel

INTERVENTIONS:
Drug: Lapatinib
  Other Names: Tyverb; Tykerb
Drug: Trastuzumab
  Other Names: Herceptin; Herclon
Drug: Endocrine Therapy — Letrozole or tamoxifen will be prescribed according to patient's menopausal status
  Other Names: Letrozol, Letrozole, Devazol, Femara, Galdar, Loxifan; Tamoxifen, Tamoxifeno, Nolvadex, Istubal, Valodex
  Arms: Dual HER2 blockade plus endocrine therapy
Drug: Paclitaxel — Only administrated if tumor progression is observed by US on week 6
  Other Names: Abraxane; Taxol

SUMMARY:
Non-randomized, open label, multicentric translational research study in women with untreated invasive breast carcinoma eligible for primary surgery (Stage I-IIIA).

The aim of PAMELA is to test the hypothesis that PAM50 HER2-enriched (HER2-E) subtype better predicts response to neoadjuvant dual anti-HER2 blockade, with or without endocrine therapy, compared to traditional clinical HER2 classification. Furthermore, we posit that characterization of gene expression patterns may identify profiles of those who may be safely spared chemotherapy.

DETAILED DESCRIPTION:
PAMELA is a non-randomized, open label, multicentric translational research study of neoadjuvant dual HER2 blockade therapy without chemotherapy. Although efficacy and safety will be investigated, the primary goal is to identify profiles predictive of clinical benefit from targeted therapy. Eligible patients must be women with untreated primary HER2-overexpressing and/or amplified breast tumors of more than 1 cm in diameter amenable to definitive surgery (stage I-IIIA).

The PAMELA study is designed to test the hypothesis that the PAM50 HER2-E subtype is able to predict clinical response to neoadjuvant dual HER2 blockade with lapatinib and trastuzumab, with or without endocrine therapy, assessed by pathological complete response in the breast (pCRB) rate at the time of surgery, compared to traditional clinical HER2 classification. Furthermore, we posit that characterization of gene expression patterns may identify profiles of those who may be safely spared chemotherapy.

Patients will first undergo screening, tumor measurement, and mandatory collection of core tumor biopsies for central determination of HER2 and HR status. These biopsies will be used to determine gene expression patterns once the patient is included in the study. Patients will be treated with dual HER2 blockade consisting of lapatinib and trastuzumab for a total of 18 weeks. Patients who are HR-positive will also be given endocrine therapy, letrozole or tamoxifen depending on their menopausal status, for the same 18 weeks. If tumor progression is observed by ultrasound (US) at week 6, tumors will be identified as resistant, and paclitaxel will be added to dual HER2 blockade, maintaining trastuzumab at the same original dose and reducing lapatinib dose for safety reasons. In those patients with HR-positive disease, endocrine therapy will be withdrawn in order to avoid its adverse interactions with chemotherapy.

Two weeks after the first administration of study medication, all patients will undergo mandatory repeat tumor tissue acquisition that will be used for secondary endpoint assessment.

Post treatment tissue acquisition will be obtained at the time of surgery from the specimen excised.

US of the breast and axillary lymph nodes will be performed at baseline, Day 14, week 6, and prior to surgery, and will be correlated with pCR. If tumor progression is observed on week 6, the US will be repeated on week 10 to discard the progression continues despite the addition of paclitaxel at neoadjuvant regimen.

Mammography is required at baseline and prior to surgery, but will not be used for the objective response assessment.

Treatment will be given until definitive surgery, clinical signs of disease progression after paclitaxel addition, unacceptable toxicity or withdrawal of patient consent.

Breast surgery will be carried out 1 to 3 weeks after completion of dual HER2 blockade with or without endocrine therapy, and 2 to 3 weeks after completion of paclitaxel plus dual HER2 blockade, should it had been initiated for progressive disease.

Following surgical excision, adjuvant treatment will be as per investigator´s choice and local standards of care outside the scope of this protocol.

End of study is 30 days (±14 days) after surgery with a safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to beginning specific protocol procedures
* Untreated invasive breast carcinoma eligible for primary definitive surgery (stage I-IIIA)
* Histologically confirmed invasive breast carcinoma, with all of the following characteristics: primary tumor ≥1 cm in largest diameter, cN0-2, No evidence of distant metastasis (M0)
* HER2-positive invasive breast cancer by central assessment, defined by ASCO/CAP guidelines
* Female patients
* Age ≥18 years
* ECOG performance status of 0 or 1
* Adequate organ function defined as: Absolute neutrophil count (ANC) ≥1.5 × 109/L, Hemoglobin (Hgb) ≥10 g/dL, Platelets >100 000/mm3, Creatinine ≤1.6 mg/dL, ALT and AST ≤2.5 × ULN, Alkaline phosphatase ≤5 ULN, Total bilirubin ≤1.5 mg/dL, Baseline LVEF ≥50% measured by echocardiography (ECHO) or Multiple Gate Acquisition (MUGA) scan
* Negative β-HCG pregnancy test (serum) for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after the menopause. All subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control from 2 weeks before administration of the first dose of investigational product until 28 days after last dose of investigational product
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* In the case of multifocal tumor (defined as the presence of two or more tumor foci in the same quadrant of the breast), the largest lesion must be ≥ 1 cm, and "target lesion" must be designated for all subsequent tumor assessments. In all tumor foci should be documented HER2 status as positive
* Availability of enough tumor sample or possibility to take a new biopsy for PAM50 analysis

Exclusion Criteria:

* Stage III inoperable breast cancer or known metastatic disease
* Patients for whom upfront chemotherapy including taxanes and anthracyclines is clinically judged appropriate as optimal neoadjuvant treatment
* Prior chemotherapy, radiotherapy or surgery for invasive breast cancer, other than excision of tumor in the contralateral breast, and provided that the patient did not previously receive adjuvant radiotherapy or chemotherapy
* Subjects with a concurrently active second malignancy, other than adequately treated non-melanoma skin cancers, in situ melanoma or in situ cervical cancer. Subjects with other non-mammary malignancies must have been disease-free for at least 5 years
* Known or suspected hypersensitivity reaction to any investigational or therapeutic compound or their incorporated substances
* Concurrent congestive heart failure or LVEF <50%
* Clinically significant (i.e. active) cardiovascular disease, including cerebrovascular accident (<6 months before enrollment), unstable angina pectoris, myocardial infarction ≤6 months before enrollment, uncontrolled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg) or high-risk uncontrolled arrhythmias
* Uncontrolled diabetes mellitus, active peptic ulcer disease or uncontrolled epilepsy
* Active uncontrolled infection at the time of enrollment
* History of significant comorbidities that, in the judgment of the investigator, may interfere with the conduction of the study, the evaluation of response, or with informed consent
* Use of any investigational agent or participation in another therapeutic clinical trial concurrently or in the previous 30 days before the enrollment
* Patients who are pregnant or breast-feeding
* Women of child-bearing potential who are unable or unwilling to use contraceptive measures
* Inability or unwillingness to abide by the study protocol or cooperate fully with the investigator
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded
* Concurrent neoadjuvant cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy other than the trial therapies)
* Concomitant use of CYP3A4 inhibitors or inducers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
pCRB to dual HER2 blockade with lapatinib and trastuzumab in all patients, at the time of surgery, predicted by PAM50 HER2-E subtype | At the time of surgery
  Comparison between the PAM50 HER2-E versus non HER2-E cases to achieve pCRB from dual HER2 blockade with lapatinib and trastuzumab at the time of surgery

SECONDARY OUTCOMES:
Pathological complete response in the breast and axilla (pCRBL) to dual HER2 blockade with lapatinib and trastuzumab, in all patients, at the time of surgery, predicted by PAM50 HER2-E subtype | At the time of surgery
  Comparison between the PAM50 HER2-E versus non HER2-E cases to achieve pCRBL from dual HER2 blockade with lapatinib and trastuzumab at the time of surgery
Residual cancer burden in the breast (RCB) to dual HER2 blockade with lapatinib and trastuzumab, in all patients, at the time of surgery, predicted by PAM50 HER2-E subtype | At the time of surgery
  Correlation between PAM50 HER2-E cases and RCB status (0-I versus II-III) after dual HER2 blockade with lapatinib and trastuzumab at the time of surgery
Changes in the percentage of Ki67-positive cells in PAM50 non-Luminal A/B (combined) subtypes | Day 14
  Comparison of the changes in the percentage of Ki67-positive cells in Luminal versus non-Luminal subtypes after 14 days of dual HER2 blockade plus endocrine therapy
Gene expression variations in all patients, in HR-negative and in HR-positive patients | Day 14
  Compare significant changes in gene expression from baseline to Day 14 in the entire study population and separately, in the HR-negative and HR-positive patients
Correlation between PAM50 HER2-E centroid, as a continuous variable, and pCR and/or RCB in the breast to dual HER2 blockade with lapatinib and trastuzumab at the time of surgery | At the time of surgery
Identification of additional gene expression signatures beyond the PAM50 subtypes that predict pCR and/or RCB to dual HER2 blockade with lapatinib and trastuzumab at the time of surgery | At the time of surgery
  In all patients and in those with HR-positive and HR-negative disease
PAM50 risk of relapse (ROR) score and its ability to predict pCR and/or RCB in the breast to dual HER2 blockade with lapatinib and trastuzumab at the time of surgery in all patients and in those with HR-positive and HR-negative disease | At the time of surgery
  Correlation between the PAM50 ROR and pCR and/or RCB after dual HER2 blockade with lapatinib and trastuzumab at the time of surgery
PAM50 HER-2 subtype (PAM50 HER2-E signature) ability as a continuous variable to predict pCRB to dual HER2 blockade at the time of surgery in patients with HR-positive disease and in patients with HR-negative disease | At the time of surgery
Changes in gene expression from day 0 to day 14, after dual HER2 blockade, that predict pCRB in all patients and in those with HR-positive and HR-negative disease | Day 14
  Identification of gene expression changes that correlate with pCRB or RCB after dual HER2 blockade treatment
Frequency of adverse events (AE) when lapatinib plus trastuzumab, with or without endocrine therapy, is administered in the neoadjuvant setting | 30 days (+/-14 days) after the surgery
  Frequency of adverse events (AE)(assessed by CTCAE v.4.03), including the following parameters:
  * All reported AEs and serious AEs
  * Neutropenia Grade 3/4
  * Febrile neutropenia Grade 3/4
  * Neuropathy Grade 3/4
  * Myalgia/arthralgia
  * Cardiotoxicity (Grade 3/4 or NYHA Class III or IV)
  * Frequency of dose reductions and dose delays due to treatment toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, MD, PhD, Study Chair — Hospital Arnau de Vilanova de Valencia; Aleix Prat, MD, PhD, Study Chair — Vall d'Hebron Institute of Oncology (VHIO); Javier Cortés, MD, PhD, Study Chair — Vall d'Hebron University Hospital
Locations (22):
- Spain (22):
  - Hospital de Torrevieja, Torrevieja, Alicante
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Institut Català d'Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital Luis Alcanyís de Xàtiva, Xàtiva, Valencia
  - Hospital Universitario Infanta Cristina, Badajoz
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Instituto Dexeus, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Arnau de Vilanova de Valencia, Valencia

REFERENCES:
- [Background] Baselga J, Bradbury I, Eidtmann H, Di Cosimo S, de Azambuja E, Aura C, Gomez H, Dinh P, Fauria K, Van Dooren V, Aktan G, Goldhirsch A, Chang TW, Horvath Z, Coccia-Portugal M, Domont J, Tseng LM, Kunz G, Sohn JH, Semiglazov V, Lerzo G, Palacova M, Probachai V, Pusztai L, Untch M, Gelber RD, Piccart-Gebhart M; NeoALTTO Study Team. Lapatinib with trastuzumab for HER2-positive early breast cancer (NeoALTTO): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2012 Feb 18;379(9816):633-40. doi: 10.1016/S0140-6736(11)61847-3. Epub 2012 Jan 17. PMID 22257673
- [Background] Gianni L, Pienkowski T, Im YH, Roman L, Tseng LM, Liu MC, Lluch A, Staroslawska E, de la Haba-Rodriguez J, Im SA, Pedrini JL, Poirier B, Morandi P, Semiglazov V, Srimuninnimit V, Bianchi G, Szado T, Ratnayake J, Ross G, Valagussa P. Efficacy and safety of neoadjuvant pertuzumab and trastuzumab in women with locally advanced, inflammatory, or early HER2-positive breast cancer (NeoSphere): a randomised multicentre, open-label, phase 2 trial. Lancet Oncol. 2012 Jan;13(1):25-32. doi: 10.1016/S1470-2045(11)70336-9. Epub 2011 Dec 6. PMID 22153890
- [Background] Prat A, Parker JS, Fan C, Perou CM. PAM50 assay and the three-gene model for identifying the major and clinically relevant molecular subtypes of breast cancer. Breast Cancer Res Treat. 2012 Aug;135(1):301-6. doi: 10.1007/s10549-012-2143-0. Epub 2012 Jul 3. PMID 22752290
- [Background] Rimawi MF, Mayer IA, Forero A, Nanda R, Goetz MP, Rodriguez AA, Pavlick AC, Wang T, Hilsenbeck SG, Gutierrez C, Schiff R, Osborne CK, Chang JC. Multicenter phase II study of neoadjuvant lapatinib and trastuzumab with hormonal therapy and without chemotherapy in patients with human epidermal growth factor receptor 2-overexpressing breast cancer: TBCRC 006. J Clin Oncol. 2013 May 10;31(14):1726-31. doi: 10.1200/JCO.2012.44.8027. Epub 2013 Apr 8. PMID 23569315
- [Background] Cancer Genome Atlas Network. Comprehensive molecular portraits of human breast tumours. Nature. 2012 Oct 4;490(7418):61-70. doi: 10.1038/nature11412. Epub 2012 Sep 23. PMID 23000897
- [Derived] Nuciforo P, Pascual T, Cortes J, Llombart-Cussac A, Fasani R, Pare L, Oliveira M, Galvan P, Martinez N, Bermejo B, Vidal M, Pernas S, Lopez R, Munoz M, Garau I, Manso L, Alarcon J, Martinez E, Rodrik-Outmezguine V, Brase JC, Villagrasa P, Prat A, Holgado E. A predictive model of pathologic response based on tumor cellularity and tumor-infiltrating lymphocytes (CelTIL) in HER2-positive breast cancer treated with chemo-free dual HER2 blockade. Ann Oncol. 2018 Jan 1;29(1):170-177. doi: 10.1093/annonc/mdx647. PMID 29045543
- [Derived] Llombart-Cussac A, Cortes J, Pare L, Galvan P, Bermejo B, Martinez N, Vidal M, Pernas S, Lopez R, Munoz M, Nuciforo P, Morales S, Oliveira M, de la Pena L, Pelaez A, Prat A. HER2-enriched subtype as a predictor of pathological complete response following trastuzumab and lapatinib without chemotherapy in early-stage HER2-positive breast cancer (PAMELA): an open-label, single-group, multicentre, phase 2 trial. Lancet Oncol. 2017 Apr;18(4):545-554. doi: 10.1016/S1470-2045(17)30021-9. Epub 2017 Feb 24. PMID 28238593
- See also: SOLTI is a non-profit academic research organization dedicated to conducting innovative breast cancer clinical trials. — http://www.gruposolti.org